CLINICAL TRIAL: NCT05566353
Title: Evaluation of the Changes in Cochlear Implant Patients Care Pathway With the Use of Telemonitoring
Brief Title: Telemonitoring in Cochlear Implant Patient Care
Acronym: EMPSICOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Toulouse (Other); Groupement Interrégional de Recherche Clinique et d'Innovation (Other); Foundation maladies rares, France (Unknown); Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL21_0519
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Hearing Loss
Keywords: Remote monitoring; Cochlear implant; Telemedicine; Healthcare system
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients followed at the implantation reference centers (Experimental): Patients eligible for implant processor renewal in 2 years and corresponding to inclusion criteria will be enrolled during their routine check-up appointment at the implantation reference centers of the University Hospitals of Montpellier and Toulouse. Patients will be their own controls through the use of their medical history data.
  Interventions: Other: Remote Check

INTERVENTIONS:
Other: Remote Check — Remote Check is a remote monitoring tool which permits patients with Cochlear Nucleus CP1000 or CP1150 processors to complete hearing tests (pure-tone and speech-in-voice audiometry, electrode impedance measures, implant functioning assessment) at home,

SUMMARY:
Following a sufficient delay after the cochlear implantation and initial implant activation, the patient will return to the hospital for follow-up visits for equipment maintenance and auditory performance evaluation only once per year. This frequency might appear either insufficient, in which case an additional patient check-up will be arranged, or excessive if patient performances and implant adjustments are stable. Using at-home testing tool for remote hearing performance monitoring can thus appear advantageous for both patients and clinicians, allowing to avoid an unnecessary journey to the implantation reference center for the first and to diminish a number of unscheduled medical appointments for the second.

DETAILED DESCRIPTION:
In December 2020, the French Medical Device and Health Technology Evaluation Committee (CNEDiMTS) voted in favour of the integration of telemonitoring in cochlear implant users' follow-up thus adding a range of new possibilities to a standard health care routine.

According to the official recommendations of the French National Authority for Health, a patient implanted for a sufficiently long time should be seen annually at the implantation reference center. This periodicity might appear too low, in which case a patient will have to organise an unscheduled check-up appointment. Such appointments are a source of various problems: firstly, they disorganise the routine of the reference centers not adapted for emergency and semi-emergency situations; secondly, the patient might encounter substantial travelling fees (only 22 refence centers in France), especially if an implant component to replace is out of stock. Having an utility of remote patient monitoring is also beneficial in situations where the access to health care system is restricted, for example, the recent pandemic of Covid 19.

Cochlear™ has recently designed an at-home based patient testing tool, Remote Check application, permitting to complete a series of hearing test from a compatible smartphone. The results are then sent to the implantation reference center and evaluated by healthcare professionals. The data is securely stored on Cloud accessible to authorised clinicians via MyCochlear site.

Although the feasibility and the accuracy in detecting technical problems of remote follow-up of people with cochlear implant had been already assessed, its impact on health care system is still unknown. Hence, this project will be the first to evaluate an interest of implementing remote monitoring in following adults with cochlear implantation.

The main objective of the study is - to determine if the use of telemonitoring through Remote Check application reduces significantly a number of unscheduled check-up appointments in the reference centre during 1 year follow-up period for a patient with a cochlear implant Cochlear™ in comparison to traditional health care approach.

The secondary objectives are:

* To compare a number of scheduled appointments during a period of Remote Check use versus a historical period of a traditional follow-up
* To compare a number of indispensable unscheduled visits (unavoidable with or without Remote Check use) with a number of unnecessary ones (avoidable with Remote Check)
* To measure the compliance of the Remote Check application use
* To assess quantitatively and qualitatively a number of implant failures/dysfunctions identified with Remote Check
* To evaluate for each study participant time spent by clinician to treat Remote Check analysis data uploaded to My Cochlear data base
* To assess patients satisfaction of Remote Check implementation in their healthcare routine
* To evaluate the quality of life specific to the Deaf before and after Remote Check use The study implies four visits for each patient. The inclusion visit (V0) is a routine check-up appointment in the implantation reference center. After the patient is informed and his/her consent is collected, the Remote Check application will be activated on his/her processor. Two next follow-up visits, V1 (V0+ 5 mois (± 0.5 mois)) and V2 (V0 + 11 mois (± 0.5 mois)), are remote visits with hearing test performed through Remote Check application. Final visit, V3 (V0 + 12 mois (± 0.5 mois)), corresponds to patient's annual check-up appointment. In case a problem with processor's functioning is detected during V2, it will be resolved at V3. Equipment verification will be also performed to detect failures missed by Remote Check.

ELIGIBILITY:
Inclusion Criteria:

* Subjects-users of uni- or bilateral cochlear implants (Cl24RE, series 400, 500 and 600) and Cochlear Nucleus processor CP1000 or CP1150 during one year minimum
* Subjects who have already renewed their processor at least once
* Subjects implanted for more than 5 years
* Over 20 years old
* Subjects with Apple or Android smartphones compatible with Remote Check

Exclusion criteria:

* Associated physical (visual, motor...) or severe cognitive (dementia, specific language development troubles) making impossible the use of smartphone software and the conduction of hearing tests
* Patients unable to give oral informed consent
* Patients residing in geographical zones with limited internet access
* Subjects deprived of liberty by juridical or administrative decision
* Patients subjected to legal protection measures (guardianship or curatorship)
* Subjects for whom French is not a native language

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Patients with at least one unscheduled follow-up visit | 24 months from the start of the study
  Annual percentage of patients-cochlear implant users having at least one unscheduled appointment at the reference center

SECONDARY OUTCOMES:
Scheduled and unscheduled visits during 1 year | 24 months from the start of the study
  The number of scheduled and unscheduled (avoidable and unavoidable) visits during 1 year
Compliance measures | 24 months from the start of the study
  The compliance will be measured by the number of Remote Check assessments in one year after the start of remote monitoring. Assessments performed within the timeframe and after the deadline will be identified.
Equipment failures and dysfunctions | 24 months from the start of the study
  The number and the type of failures/dysfunctions identified by Remote Check
Time spent in MyCochlear for each patient | 24 months from the start of the study
  Clinician login time spent on each subject's file on MyCochlear data base during the year of follow up
Patient satisfaction | 24 months from the start of the study
  Patient satisfaction measured by the questionnaire validated in French language: "the Service User Technology Acceptability (SUTAQ)". Score will be assessed by 5 options from "Strongly disagree" (worse outcome), "Disagree somewhat", "Neither agree nor disagree", "agree somewhat" to "strongly agree" (better outcome)
Patient's Quality of Life | 24 months from the start of the study
  Patient's quality of life score linked to deafness will be measured by the questionnaire Speech, Spatial and Qualities of Hearing scale (Sp-SSQ12) validated in french. Score will run from 0 (worse outcome) to 10 (better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided